CLINICAL TRIAL: NCT03911804
Title: The Effect of Continuous Epidural Analgesia on Intracranial Pressure by Measuring the Optic Nerve Sheath Diameter Using Ultrasound in Pediatric Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1-2019-0004
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Osteotomy of Lower Extremity
MeSH Terms: interventions — Anesthesia, Epidural

STUDY DESIGN:
Intervention Model Description: Randomly selected patients of the bolus group are given 0.3 ml/kg bolus/hr of 0.15% ropivacaine for epidural analgesia. In contrast, patients in the infusion group are given 0.3 ml/kg/hr 0.15% ropivacaine at a constant rate for epidural analgesia.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants, care providers and investigators are blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bolus group (Experimental)
  Interventions: Procedure: bolus group and infusion group for epidural block
- Infusion group (Active Comparator)
  Interventions: Procedure: bolus group and infusion group for epidural block

INTERVENTIONS:
Procedure: bolus group and infusion group for epidural block — Randomly selected patients of the bolus group are given 0.3 ml/kg bolus/hr of 0.15% ropivacaine for epidural analgesia. In contrast, patients in the infusion group are administered 0.3 ml/kg/hr 0.15% ropivacaine at a constant rate for epidural analgesia.

SUMMARY:
Ultrasonography of optic nerve sheath diameter shows a good level of diagnostic accuracy for detecting intracranial hypertension. The aim of this study is to evaluate the effect of continuous epidural block on intracranial pressure in pediatric patients undergoing osteotomy of lower extremity. Forty patients, aged 4 years to 13 years, receiving epidural analgesia before osteotomy will be divided into bolus group (n=30) and infusion group (n=30). Randomly selected patients of the bolus group are given 0.3 ml/kg bolus/hr of 0.15% ropivacaine for epidural analgesia. In contrast, patients in the infusion group are administered 0.3 ml/kg/hr 0.15% ropivacaine at a constant rate for epidural analgesia. The primary endpoint is the difference in the optic nerve sheath diameter after epidural analgesia measured by optic nerve ultrasonography between groups.

ELIGIBILITY:
Inclusion Criteria:

* 1. Pediatric patients from 4 to 13 years of age undergoing osteotomy of lower extremity

Exclusion Criteria:

* 1. Patients with contraindications to epidural analgesia (local infection, clotting disorders, anatomical abnormalities, sepsis, etc.)
* 2. Patients with symptoms or signs associated with a history of elevated intracranial pressure or elevated intracranial pressure
* 3. Patients with ophthalmic disease or surgery
* 4. The estimated operation time is less than 180 minutes.
* 5. All parents of the subject are foreigners or illiterate

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
The difference in the optic nerve sheath diameter (ONSD) between groups | Before epidural block
  The optic nerve sheath diameter measured by optic nerve ultrasonography
The difference in the optic nerve sheath diameter (ONSD) between groups | 30 minutes after epidural block
  The optic nerve sheath diameter measured by optic nerve ultrasonography
The difference in the optic nerve sheath diameter (ONSD) between groups | 60 minutes after epidural block
  The optic nerve sheath diameter measured by optic nerve ultrasonography
The difference in the optic nerve sheath diameter (ONSD) between groups | 90 minutes after epidural block
  The optic nerve sheath diameter measured by optic nerve ultrasonography
The difference in the optic nerve sheath diameter (ONSD) between groups | 120 minutes after epidural block
  The optic nerve sheath diameter measured by optic nerve ultrasonography
The difference in the optic nerve sheath diameter (ONSD) between groups | 180 minutes after epidural block
  The optic nerve sheath diameter measured by optic nerve ultrasonography

SECONDARY OUTCOMES:
The difference in the number of patients whose ONSD values increased to more than 5.75 mm at each time point between the two groups | Before epidural block
  The optic nerve sheath diameter measured by optic nerve ultrasonography
The difference in the number of patients whose ONSD values increased to more than 5.75 mm at each time point between the two groups | 30 minutes after epidural block
  The optic nerve sheath diameter measured by optic nerve ultrasonography
The difference in the number of patients whose ONSD values increased to more than 5.75 mm at each time point between the two groups | 60 minutes after epidural block
  The optic nerve sheath diameter measured by optic nerve ultrasonography
The difference in the number of patients whose ONSD values increased to more than 5.75 mm at each time point between the two groups | 90 minutes after epidural block
  The optic nerve sheath diameter measured by optic nerve ultrasonography
The difference in the number of patients whose ONSD values increased to more than 5.75 mm at each time point between the two groups | 120 minutes after epidural block
  The optic nerve sheath diameter measured by optic nerve ultrasonography
The difference in the number of patients whose ONSD values increased to more than 5.75 mm at each time point between the two groups | 180 minutes after epidural block
  The optic nerve sheath diameter measured by optic nerve ultrasonography

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Lin Y, Li Q, Liu J, Yang R, Liu J. Comparison of continuous epidural infusion and programmed intermittent epidural bolus in labor analgesia. Ther Clin Risk Manag. 2016 Jul 14;12:1107-12. doi: 10.2147/TCRM.S106021. eCollection 2016. PMID 27471390
- [Background] Padayachy LC, Padayachy V, Galal U, Pollock T, Fieggen AG. The relationship between transorbital ultrasound measurement of the optic nerve sheath diameter (ONSD) and invasively measured ICP in children. : Part II: age-related ONSD cut-off values and patency of the anterior fontanelle. Childs Nerv Syst. 2016 Oct;32(10):1779-85. doi: 10.1007/s00381-016-3068-4. Epub 2016 Sep 20. PMID 27659820